CLINICAL TRIAL: NCT01373632
Title: Multicenter, Randomized, Non-inferiority Study of Firebird 2 Versus Excel Sirolimus-eluting Stent in Treating Real-world Patients With Coronary Artery Disease
Brief Title: Firebird 2 Versus Excel Sirolimus-eluting Stent in Treating Real-world Patients With Coronary Artery Disease
Acronym: FESTA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Cardiovascular Department
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20110611
Record Dates: First submitted 2011-06-13; First posted 2011-06-15 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Coronary Artery Disease
Keywords: significant stenosis (>70% of lumen stenosis); epicardial coronary arteries; clinical ischemic
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Firebird 2 stent group (Experimental): the patients who receive Firebird 2 stent
  Interventions: Device: Firebird 2 sirolimus-eluting stent
- Excel stent group (Active Comparator): the patients who receive Excel stent
  Interventions: Device: Excel sirolimus-eluting stent

INTERVENTIONS:
Device: Firebird 2 sirolimus-eluting stent — the Firebird 2 sirolimus-eluting stent is a SES with durable polymer based on Co-Cr stent platform
  Arms: Firebird 2 stent group
Device: Excel sirolimus-eluting stent — the Excel sirolimus-eluting stent is a stent with biodegradable polymer (PLA) based on stainless steel (316L) stent platform
  Arms: Excel stent group

SUMMARY:
Sirolimus-eluting stent (SES) has been world-widely used in clinical practice in treating patients with coronary artery disease (CAD). The efficacy and safety of Excel SES (JW Medical, Shandong, China, MA) with biodegradable polymer has been proved by several clinical trials. Here the investigators design a prospective, multicenter, randomized clinical study in purpose of identifying the non-inferiority in the efficacy and safety in treating CAD patients by Firebird 2 SES (Microport, Shanghai) with durable polymer, comparing with Excel SES.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* male or un-pregnant female
* stenosis > 70% in one of major the epicardial coronary arteries
* no contra-indications of stent implantation
* singed the informed consent

Exclusion Criteria:

* acute myocardial infarction within one week
* have contra-indications of stent implantation or can not tolerate dual antiplatelet therapy
* no history of stent implantation within last one-year
* received other brand coronary stent during index procedure
* with no achievement of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-06 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
in-stent late lumen loss at 9 months' angiographic follow-up | 9 months
  patients are planned to receive angiographic follow-up at 9 months after index procedure, and in-stent late lumen loss will be analyzed

SECONDARY OUTCOMES:
target vessel failure | 2 years after index procedure
  defined as the occurrence of any of the following within 1 and 2 years after the index procedure: death from cardiac causes, Q-wave or non-Q-wave myocardial infarction, or revascularizationof the target vessel (emergency or elective coronaryartery bypass grafting [CABG] or repeated percutaneous transluminal coronary angioplasty [PTCA]).

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Zhang Q, Xu B, Yang YJ, Zhang RY, Li JP, Qiao SB, Zhang JS, Hu J, Qin XW, Hong T, Chen JL, Huo Y, Shen WF, Gao RL. Sirolimus-eluting cobalt alloyed stents in treating patients with coronary artery disease: six-month angiographic and one-year clinical follow-up result. A prospective, historically controlled, multi-center clinical study. Chin Med J (Engl). 2007 Apr 5;120(7):533-8. PMID 17442198
- [Background] Han Y, Jing Q, Chen X, Wang S, Ma Y, Liu H, Luan B, Wang G, Li Y, Wang Z, Wang D, Xu B, Gao R. Long-term clinical, angiographic, and intravascular ultrasound outcomes of biodegradable polymer-coated sirolimus-eluting stents. Catheter Cardiovasc Interv. 2008 Aug 1;72(2):177-83. doi: 10.1002/ccd.21600. PMID 18655114